CLINICAL TRIAL: NCT01464385
Title: Nutrition Beverage Tolerance Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BK98
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Human Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nutritional Beverage #2 (Experimental): Nutritional Beverage with an amino acid Oral 237 ml
  Interventions: Other: Nutritional Beverage
- Nutritional Beverage #3 (Experimental): Nutritional Beverage with an amino acid Oral 237 ml
  Interventions: Other: Nutritional Beverage
- Nutritional Beverage #1 (Placebo Comparator): Nutritional Beverage Oral 237 ml
  Interventions: Other: Nutritional Beverage

INTERVENTIONS:
Other: Nutritional Beverage — Nutritional Beverage Oral 237mL
  Arms: Nutritional Beverage #1
Other: Nutritional Beverage — Nutritional Beverage Oral 237 mL
  Arms: Nutritional Beverage #2
Other: Nutritional Beverage — Nutritional Beverage Oral 237mL
  Arms: Nutritional Beverage #3

SUMMARY:
To evaluate the sensations experienced by subjects consuming a nutritional beverage.

ELIGIBILITY:
Inclusion Criteria:

Subject ≥ 45 years of age.

If female, subject is either postmenopausal for at least 1 year or surgically sterile

Subject reports that he/she has not participated in a research study in the last three months.

Exclusion Criteria:

Subject has active metabolic or endocrine disease

Subject has an autoimmune disorder

Subject has a disorder of gastrointestinal tract or any gastrointestinal surgery in past 12 months.

Subject has food allergy, celiac disease or intolerance to any of the ingredients in the study products

Subject reports history of parasthesia; and/or is currently taking medication/dietary supplements/substances that may cause parasthesia for 4 weeks prior to screening

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects experiencing neurologic adverse event(s) | 2-3 weeks

SECONDARY OUTCOMES:
Proportion of subjects experiencing any adverse event(s). | 2-3 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Chair — Abbott
Locations (1):
- The National Food Lab, Livermore, California, United States